CLINICAL TRIAL: NCT03413722
Title: Alterations in Cognitive Function and Cerebral Blood Flow After Conversion From Calcineurin Inhibitors to Everolimus
Brief Title: Alterations in Cognitive Function and Cerebral Blood Flow After Conversion From Calcineurin Inhibitors (CNIs) to Everolimus
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Aditi Gupta, MD, Associate Professor, University of Kansas Medical Center
Other Study IDs: STUDY00140594; CRAD001AUS211T (Other Grant/Funding Number: Novartis Pharmaceuticals)
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: End Stage Renal Disease
Keywords: Kidney transplant; Cognitive function
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus; Everolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conversion Group: Kidney transplant recipients at the University of Kansas Medical Center (KUMC) who are currently on tacrolimus (CNI), and will be undergoing conversion to Everolimus + low dose CNI. Potential participants will be asked to participate in the study after the decision to convert CNI to Everolimus + low dose CNI has been made.
  Interventions: Drug: Tacrolimus; Drug: Everolimus
- Control Group: Kidney transplant recipients at KUMC on tacrolimus (CNI). These will be patients not planning to undergo any change in immunosuppression.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — The patient's physician will prescribe drug according to standard practice.
  Other Names: Prograf
Drug: Everolimus — The patient's physician will prescribe drug according to standard practice.
  Groups: Conversion Group

SUMMARY:
The purpose of this study is to learn if changing from Tacrolimus to Everolimus will improve cognitive function by having less effect on brain blood flow.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* able to sign informed consent
* able to arrange transportation to and from study site
* without acute stroke, concussion or traumatic brain injury
* without acute medical issues at the time of participation
* At least 12 weeks post Kidney transplant surgery

Exclusion Criteria:

* are claustrophobic or have other contra-indication for magnetic resonance imaging (MRI)
* have hearing or visual impairment
* are unable to read, write, speak or understand English
* have uncontrolled psychosis or seizure disorder or are currently using antipsychotics or anti-epileptics
* taking Envarsus at the time of recruitment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be patients undergoing kidney transplant at the University of Kansas Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | Change from Baseline to Week 12

SECONDARY OUTCOMES:
Change in cerebral blood flow | Change from Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Gupta, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States